CLINICAL TRIAL: NCT06537193
Title: A Prospective Multicenter Study for the Intra-Individual Comparison of Abbreviated MRI Using Gadoxetic Acid and Dynamic CT for Surveillance of Recurrent HCC After Curative Treatment
Brief Title: Abbreviated MRI Using Gadoxetic Acid Versus CT for Surveillance of Recurrent HCC After Curative Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-1630
Record Dates: First submitted 2024-07-30; First posted 2024-08-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Abbreviated MRI; Dynamic CT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMRI and CT (Experimental): Procedure: AMRI examination The study subjects will receive intravenous injection of gadoxetic acid (0.025 mmol/kg, Primovist; Bayer, Berlin, Germany) in the waiting room and then proceed to the examination room for MRI testing 15-20 minutes later. The MRI examination will be conducted using a 3-Tesla MRI machine, and the MRI protocol will consist of T2-weighted imaging, diffusion-weighted imaging (b value of 0, 50, and 500 s/mm2), and hepatobiliary phase imaging.
  Procedure: dynamic CT CT will be performed by obtaining dynamic phases (precontrast phase, arterial phase, portal venous phase, and delayed phase images). Subjects will receive intravenous injection of iodine contrast media. Scan coverage will be from the basal lung to the iliac crest or pelvis.
  Interventions: Diagnostic Test: AMRI; Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: AMRI — The study subjects will receive intravenous injection of gadoxetic acid (0.025 mmol/kg, Primovist; Bayer, Berlin, Germany) in the waiting room and then proceed to the examination room for MRI testing 15-20 minutes later. The MRI examination will be conducted using a 3-Tesla MRI machine, and the MRI protocol consists of T2-weighted imaging,diffusion-weighted imaging (b value of 0, 50, and 500 s/mm2), and hepatobiliary phase imaging.
Diagnostic Test: CT — CT will be performed by obtaining dynamic phases (precontrast phase, arterial phase, portal venous phase, and delayed phase images). Subjects will receive intravenous injection of iodine contrast media. Scan coverage was from the basal lung to the iliac crest or pelvis.

SUMMARY:
Hepatocellular carcinoma (HCC) often has a poor prognosis after curative treatment due to frequent recurrence. Post-surgery, 60-70% of HCC patients experience recurrence, rising to 80% after ablation therapy. This is partly because underlying cirrhosis or chronic liver disease remains, increasing the risk of secondary HCC. The risk of recurrence varies over time, with a high risk in the first two years due to micro-metastasis. Later recurrences are usually new primary cancers (de novo HCC). Therefore, regular imaging tests, such as computed tomography (CT) or magnetic resonance imaging (MRI) every three months in the first two years, are necessary for early detection, but guidelines for post-two-year screenings are unclear.

Currently, for patients recurrence-free for two years, contrast-enhanced liver CT or MRI is performed every 3-6 months as a secondary screening test. However, repeated use of CT raises concerns about radiation exposure and iodine-based contrast agents can lead to side effects and kidney issues. MRI with hepatocyte-specific agents like gadoxetic acid (Primovist) is effective but costly and time-consuming, with potential side effects from repeated gadolinium exposure. Therefore, there is a need for a validated secondary screening method that is both effective and reduces patient risk.

Abbreviated contrast-enhanced MRI, using only essential sequences, has shown promise in retrospective studies for detecting HCC. However, these studies have limitations, such as potential bias and lack of data on repeated screenings. There is limited research on secondary screening post-curative treatment for HCC. This study aims to prospectively evaluate the use of abbreviated contrast-enhanced MRI with Primovist as a secondary screening method for detecting secondary HCC in patients who have been recurrence-free for more than two years.

DETAILED DESCRIPTION:
A total of 455 subjects will be evaluated by two rounds of tests with both abbreviated MRI (AMRI) and dynamic CT to detect the occurrence of secondary HCC. These two imaging tests are planned to be performed twice, with a basic interval of 16 weeks between tests. However, considering the clinical practice of varying the imaging intervals based on the patient's risk level, the actual interval between tests can range from 4 to 8 months. If a suspicious lesion indicative of HCC is detected during the study, a recall examination using complete MRI will be performed within 3 months. If the recall examination does not confirm the diagnosis, a contrast-enhanced ultrasound or biopsy will be conducted. The diagnosis of HCC will be made based on international guidelines, with a histological confirmation or classification as Liver Imaging-Reporting and Data System (LI-RADS) category 5. After the completion of the two evaluation rounds, at least 6 months of clinical follow-up data will be collected to record the occurrence of interval cancer. If HCC is confirmed during the study, the participant will be excluded from further study participation, and the treatment will proceed according to current clinical processes. If no lesions are detected during the two surveillance rounds, follow-up for up to 6 months after the second test will be conducted according to current clinical processes. If HCC is diagnosed, which is the primary outcome of the study, the study will be considered complete, and this will not be treated as an adverse event of the study. If a patient chooses not to continue participating in the study during the repeated application of the protocol, the study for that patient will conclude, even if the two rounds of testing are not completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with more than two years without recurrence after curative treatment (surgery or local ablation) for HCC
2. Patients with no history of systemic treatment, radiation therapy, or trans-arterial chemoembolization for HCC
3. Older than 20 years of age
4. Eastern Cooperative Oncology Group performance status of 0-2
5. Patient is able to comply with scheduled visits, evaluation plans, and other study procedures
6. Patient is willing to provide written informed consent

Exclusion Criteria:

1. Active or suspected cancer, or a history of malignancy where the risk of recurrence is equal or higher than 20% within 2 years.
2. Significant medical comorbidities in which survival is predicted to be less than 3 years
3. Estimated glomerular filtration rate < 30 mL/min/1.73m²
4. Patient not eligible for applying LI-RADS criteria, such as Budd-Chiari Syndrome
5. Precautions for MRI (cardiac pacemaker, severe claustrophobia that may interfere with protocol compliance).
6. Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with completing the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate (DR) of patients with HCC | 6 months after the completion of the 2 surveillance rounds
  DR = True positive / True positive + False positive + True negative + False negative
False referral rate (FRR) of patients with HCC | 6 months after the completion of the 2 surveillance rounds
  FRR = False positive / True positive + False positive + True negative + False negative

SECONDARY OUTCOMES:
DR of patients with early stage HCC | 6 months after the completion of the 2 surveillance rounds
  DR = True positive / True positive + False positive + True negative + False negative
FRR of patients with early stage HCC | 6 months after the completion of the 2 surveillance rounds
  FRR = False positive / True positive + False positive + True negative + False negative
DR of patients with very early stage HCC | 6 months after the completion of the 2 surveillance rounds
  DR = True positive / True positive + False positive + True negative + False negative
FRR of patients with very early stage HCC | 6 months after the completion of the 2 surveillance rounds
  FRR = False positive / True positive + False positive + True negative + False negative

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu , 88, Olympic-ro 43-gil, South Korea

IPD SHARING:
Plan to Share IPD: No